CLINICAL TRIAL: NCT05974761
Title: Clinical Observation on the Treatment of Chronic Low Back Pain With Side-lying Massage Based on Fascia Chain
Brief Title: Clinical Observation on the Treatment of Massage Based on Fascia Chain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: muxing zhu (Other)
Responsible Party: Sponsor-Investigator, muxing zhu, Professor, Shandong University of Traditional Chinese Medicine
Organization: Shandong University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: jigubchao202307; Z-2022046 (Other Grant/Funding Number: Health Commission of Shandong Province)
Record Dates: First submitted 2023-07-07; First posted 2023-08-03 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Side lying muscle massage (Experimental): The patient was placed in a lateral decubitus position with the physician standing on the ventral side of the patient, with the crotch resting on the anterior edge of the superior iliac crest, and the elbow rising from the medial side of the highest point of the superior iliac crest, follow the palpation (avoiding the L3 transverse process) along the steep edge of the skeleton slowly toward the spine, and focus on the painful points or cords by repeatedly applying the elbow press method and the elbow flick method for 1-2 minutes, after that, the tendon was found to be induration with elbow tip probing, and the tendon was plucked 3-5 times vertically along the vertical direction.
  Interventions: Other: massage
- Traditional Chinese massage (Other): Through the point, massage, bone-setting treatment
  Interventions: Other: Traditional Chinese massage

INTERVENTIONS:
Other: massage — The patient was placed in a lateral decubitus position with the physician standing on the ventral side of the patient, with the crotch resting on the anterior edge of the superior iliac crest, and the elbow rising from the medial side of the highest point of the superior iliac crest, follow the palpation (avoiding the L3 transverse process) along the steep edge of the skeleton slowly toward the spine, and focus on the painful points or cords by repeatedly applying the elbow press method and the elbow flick method for 1-2 minutes, and then the elbow tip contact to find the sinew knot and along the vertical direction of 3-5 times, the force should be deep penetration.
  Arms: Side lying muscle massage
Other: Traditional Chinese massage — Through the point, massage, bone-setting treatment
  Arms: Traditional Chinese massage

SUMMARY:
The goal of thisclinical trial is to observe and quantify the impact of our massage methods on the human body based on B-mode ultrasound, Vas score, and ODI score, and to compare our massage methods with traditional Chinese massage treatment. The main questions it aims to answer are:

* To set up our standard operating procedure of massage therapy to adjust the stress line of psoas myofascial chain, and provide a more simple and effective therapy for Chronic low back pain.
* try to establish a kind of ultrasonic standard to evaluate the curative effect of treating chronic low back pain.

The subjects were randomly divided into two groups, the experimental group and the control group, the experimental group was given our characteristic massage treatment, the control group was given traditional Chinese massage treatment.Both groups were treated once every other day, 3 times a week, 2 weeks as a course of treatment, 2 courses of treatment.

DETAILED DESCRIPTION:
1. the patients in the observation group were treated with the manipulation of side-lying and tendons poking. The specific manipulation methods were as follows: (1) the relaxation method: the patients were in prone position, in order to relieve the superficial muscle and fascia, the doctor applied the method of massage, palm massage and arm movement up and down the vertical spine muscle for 3-5 minutes, move your body as close to the bedside as possible. Straighten your lower legs, bend your hips and knees, rest your ankles on your lower legs, and lift your arms to the side of your head. The surgeon stands on the ventral side of the patient, with the crotch resting on the anterior edge of the superior iliac crest, with the elbow rising from the medial top of the superior iliac crest, and slowly following the palpation along the vertical edge of the skeleton toward the spine (avoiding the L 3 transverse process) , and focus on the pain point or the rope to repeatedly apply elbow pressure, elbow plucking method 1-2 minutes to ease the spasm and analgesia, ease adhesion, promote the absorption of inflammatory edema, manipulation is appropriate to ease the gentle; Then the elbow moved down to the buttocks, with the elbow tip touch to find the sinew knot and along the vertical direction of the vertical plucking 3-5 times, the force should be deep penetration. (3) the method of adjusting the extensor muscles and bones: keeping the upper posture, doing the lumbar oblique pulling, one time each side, further stretching the deep muscles of the waist, adjusting the disorder of the lumbar facet joints caused by the twinning contraction of the muscles and fascia. 4 ending type: with double palm up and down alternately percussion waist muscle ten times to end.
2. control group: according to the Tuina treatment scheme of low back pain in the textbook of the 13th five-year plan for higher education of Chinese medicine published by China Traditional Chinese Medicine Press in July 2016 and edited by Fan Binghua. The specific methods of operation are as follows: 1 relaxation method: the patient lies prone, the operator stands on the affected side, and applies the massage to the affected side waist, arm and thigh back and forth for 5 minutes, the strength should be deep and gentle, in order to relax the tendons and activate the blood circulation, promote the absorption of peripheral inflammation and edema. 2 point method: the Doctor uses one finger to push the middle acupoints in Ashi, Shenshu, Baihuanshu, Huantiao, zhibian, Chengfu, and massages each point for about half a minute to relax the muscles and activate the blood, 3 method of relieving spasm and pain: the Doctor applied the thumb plucking method at the tendon of the cord-like muscle 2-3cm below the medial side of the highest point of the skeletal crest. The manipulation was from light to heavy, and could be alternately operated with the thumb pressing and kneading method for about 2 minutes, in order to release adhesion, Pain Relief 4 end: the operator to small thenar vertical rub both sides of the erector muscles, transverse rub lumbosacral department, diaphanous heat for the degree. To double palm up and down alternately tap the lumbosacral end of a dozen times. The Observation Group and the control group were treated once every other day, 3 times a week, 2 weeks as a course of treatment, 2 courses of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Those who met the diagnostic criteria of chronic low back pain, aged 18-65 years, volunteered to join the trial and signed the informed consent.

Exclusion Criteria:

* In the course of treatment, the skin of waist and buttocks was obviously damaged, infected and ulcerated, and the women were in the period of menstruation, pregnancy or lactation Patients with cardiac cerebrovascular disease, hepatic and renal insufficiency, bleeding disorders and mental disorders, and participants in other clinical trials within one month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-10-21 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The changes of fascia of erector spine muscle before and after 4 weeks treatment were compared. | 24months
  The position of the lower edge of the transverse process of T12, the lower edge of the transverse process of L 3 and the upper edge of the sacral pathway were determined, take these three points as the placement point of probe center position. After placing the probe, move the probe up and down to get a clear echo of the center point. The musculus erectus erectus muscle appeared between l 3 transverse process, T 12 transverse process lower edge, sacral camel upper edge and fascia layer lower edge, and the thickness of musculus erectus erectus muscle was measured in turn. 3 measurements are required at the same location, and the mean value is taken as the corrected thickness value.
The changes of Vas score were compared before and after 4 weeks treatment | 24months
  Before and after the treatment, the changes of the thickness membrane of the erector spine muscle were observed by b-mode ultrasonography, and the therapeutic effect of lateral supine massage on Psoas myofascitis was quantitatively expressed,A straight line with a ruler is divided into 10 segments, with 0 and 10 marks at both ends. The larger the scale, the higher the pain level. 0 was painless, 1-3 was mild pain that could be tolerated, 4-6 was pain that affected sleep but could be tolerated, 7-9 was pain that was gradually intense and affected appetite and sleep, and 10 was severe pain.
The changes of ODI score were compared before and after 4 weeks treatment | 24months
  Before and after the treatment, the changes of the thickness membrane of the erector spine muscle were observed by b-mode ultrasonography, and the therapeutic effect of lateral supine massage on Psoas myofascitis was quantitatively expressed,It was divided into 10 related questions, such as pain intensity, self-care ability, lifting ability, walking ability, sitting ability, walking ability, ability, standing time and sleep quality. There are 6 options for each question, with scores ranging from 0 to 5. The maximum cumulative score for 10 questions is 50. The formula is: Total Score = (score/5 × number of questions answered) × 100% . The higher the score, the more severe the dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: shuwen mao, Principal Investigator — Shandong University of Traditional Chinese Medicine
Locations (1):
- Affiliated Hospital of Shandong University of traditional Chinese medicine, Jinan, Shandong, China